CLINICAL TRIAL: NCT03940456
Title: Prognostic Factors of Importance on Who Develops Chronic Low Back Pain: A Protocol Update for an Inception Cohort With Focus on Prognostic Factors With 54 Years of Follow up
Brief Title: Prognostic Factors of Importance on Who Develops Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Other Study IDs: Elsinore low back pain cohort
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain; Life Style; Illness Perception
Keywords: Cohort; Low Back Pain; Illness perception; Life Style
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inception cohort, former Elsinore pupils: 640 former Elsinore pupils (330 female, 310 male). Aged 14 in 1965. Two earlier cross-sectional studies have been done in this group (in 1990 and 2000).
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire mainly focusing on low back pain, pain related disorders, psychosocial factors and the use of alternative treatments for pain

SUMMARY:
The incidence of low back pain (LBP) is increasing and prognostic factors for developing LBP are unclear. Based on questionnaires, different prognostic factors are being explored over time.

DETAILED DESCRIPTION:
Despite massive efforts of trying to find predictors and prevention for LBP, it remains to be clarified, why some individuals develop severely disabling low back pain while others never experience noteworthy back pain. There is no evidence that numbers of chronically affected individuals have diminished; rather, the incidence of LBP has increased continuously over the last 20 years which is also reflected in rising numbers of lumbar surgical treatments. The prevalence and burden increase with age and prevention of LBP in an aging population seems more urgent than ever. As LBP is undoubtedly a multifaceted disorder that tends to fluctuate throughout life, there is a need for longitudinal research, exploring the effect of both life style and psychosocial factors on the development of chronic low back pain.

The aim of this study is to identify whether a history of low back pain during adolescence represents an increased risk of experiencing low back pain later in life.

ELIGIBILITY:
Inclusion Criteria:

This is an inception cohort based on pupils from schools in Elsinore. There are no formal inclusion criteria other tan being part of this cohort

Exclusion Criteria:

* No formal exclusion criteria but inability to understand/answer our questionnaire is per se an exclusion criteria

Ages: 67 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Study population will comprise all available subjects who have been part of the Elsinore cohort since 1965
Sampling Method: Non-Probability Sample
Enrollment: 607 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
prevalence of LBP | measured once at study baseline
  To estimate the prevalence of self-disclosed low back pain

SECONDARY OUTCOMES:
Incidence of LBP | measured once at study baseline
  To estimate the incidence of self-disclosed low back pain
Brief illness perception questionnaire (IPQ-B) | measured once at study baseline
  Actual IPQ-B score. Generic questionnaire developed to measure illness perception. The IPQ-B contains eight items and one causal scale. Items 1-8 are rated using a 0-to-10 response scale, item 9 is a memo field. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7).
  A low score on items number 1,2,5,6 and 8 indicates that the illness is perceived as benign while a low score on the items 3, 4 and 7 indicates that the illness is perceived as threatening. By reversing these three items it is possible to compute an overall score. A higher score reflects a more threatening view of the illness.
EQ-5D (3 likert scale) | measured once at study baseline
  The EQ-5D-3L essentially consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS) (0-100). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' (100) and 'Worst imaginable health state' (0). This information can be used as a quantitative measure of health outcome as judged by the individual respondents. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided